CLINICAL TRIAL: NCT02121873
Title: The Breast Duct: Pilot Study of Genomic Sequencing of Exfoliated Ductal Cells Obtained Through Endoscopy and Lavage
Status: Completed | Type: Observational
Sponsor: Atossa Therapeutics, Inc. (Industry)
Collaborators: Covance (Industry); Illumina, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: L-503
Record Dates: First submitted 2014-04-15; First posted 2014-04-24 (Estimated); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Breast Cancer; Preneoplastic Conditions; Ductal Carcinoma in Situ
Keywords: breast cancer, nipple aspirate, ductal lavage, hyperplasia
MeSH Terms: conditions — Breast Neoplasms; Precancerous Conditions; Carcinoma, Intraductal, Noninfiltrating; Hyperplasia | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, nipple aspirate fluid, ductal lavage fluid
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women with and without breast cancer: Nipple aspirator, ductal lavage microcatheter, blood draw
  Interventions: Device: Nipple aspirator; Device: Ductal lavage microcatheter; Device: Blood draw

INTERVENTIONS:
Device: Nipple aspirator — The subject will undergo nipple aspiration with a suction device designed to elicit fluid from the nipple.
  Other Names: Forecyte breast aspirator
Device: Ductal lavage microcatheter — Upon completion of the nipple aspiration procedure, subjects will undergo a nipple block with local anesthesia. The duct will be lavaged with the ductal lavage microcatheter. Samples will be immediately processed for shipping to Covance for WGS. Subjects will be contacted 24 hours and again 2 weeks after the procedure to collect any untoward effects of participating in the study.
  Other Names: FullCYTE Microcatheter
Device: Blood draw — Blood will be drawn and immediately processed for shipping to Covance for WGS.

SUMMARY:
The objective of this study is to determine whether we can use minimally invasive techniques to gain access to exfoliated ductal epithelial cells for whole genome sequencing.

1. To examine women with nipple aspiration, ductoscopy and ductal lavage and collect exfoliated cells from two ducts per woman.
2. To collect a blood sample at the time of the examination in order to obtain the woman's baseline genomic sequence.
3. De-identified samples will then have DNA and RNA extracted and whole genome sequencing and transcriptome analysis performed by Covance and Illumina.
4. Comparisons will be made within a breast (two ducts) and between the duct and blood as well as between women.

DETAILED DESCRIPTION:
Despite the lack of anatomical clarity in the literature, Tibor Tot has postulated that breast cancer and DCIS are a lobar disease as the simultaneously or asynchronously appearing, often multiple in situ tumor foci are localized within a single "sick" lobe. This theory has some resonance in the molecular studies that have been done in the breast demonstrating that there are large "patches" of clonality even in normal breast tissue. Most of this work was based on microdissection, however, and assumes that adjacent duct profiles belong to the same lobe. In fact both Cooper and Going have shown intertwining of arborizing ducts from different independent lobes. This sets the stage for errors of interpretation in micro-dissected tissue.

Ductal lavage allows the cannulation and lavage of individual ducts and collection of 1,000- over 10,000 exfoliated cells that can be studied for molecular and genetic changes. Ductoscopy adds the ability to confirm that the duct has not been perforated and to brush the lining of the duct to increase cell yield. Real-time ultrasound can be used to confirm the ductal anatomy. With the combination of these minimally invasive techniques it is now possible to collect the cells needed to apply new genetic techniques and investigate the genome of the ductal epithelial cell.

While the methods for obtaining the ductal epithelial cells have been being developed similar advances have been made in whole genome sequencing technology. Knome®, a for-profit company, is now able to analyze ductal cells against blood to identify variants, including single nucleotide polymorphisms (SNP's), short and long insertions and deletions (indels), inversions, translocations, fusion genes and copy number variations (CNVs). Ingenuity Pathway Analysis can identify mRNA networks that can be driving pre-cancerous hyperplasia. Covance Genomics Laboratory (CAL) will perform DNA and RNA extraction, DNA QC and Next-Generation Sequencing on the Illumina platform.

With the combination of these minimally invasive techniques and Next-Generation Sequencing we will be able to test our hypothesis that it is now possible to interrogate the genetic sequence of a single normal duct and to compare it to the sequence in the blood to identify early epithelial mutations. In addition by comparing the sequence of two ducts in one breast we can gain insight into whether each duct is clonal or the whole breast shares the same genetic pattern. And finally, understanding the pathways that are activated in pre-cancerous duct lesions can provide targets for intraductal treatment programs.

ELIGIBILITY:
Inclusion Criteria:

* Be female
* Have at least one intact nipple
* If over 50, have had a normal mammogram within 12 months prior to the enrollment date
* Have a normal physical examination of the breast to be studied within 12 months prior to the enrollment date
* Be > 18 years of age
* Sign the informed consent form

Exclusion Criteria:

* Be currently pregnant or pregnant within the last 12 months
* Be currently lactating or lactated within the last 12 months
* Have received chemotherapy in the last 12 months
* Have had an abnormal mammogram within the last year
* Have had any subareolar or other surgery (papilloma resections, biopsies or fine needle aspirations) within 2 centimeters of the nipple (biopsies and fine needle aspirations >2 centimeters from the nipple are acceptable)
* Have active infections or inflammation in a breast to be studied
* Have a known allergy to lidocaine
* Be unwilling to sign informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women will be recruited from our local pool of volunteers who have participated in previous studies of ductal lavage and/or ductoscopy at the Foundation.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-07; Primary Completion 2011-09 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Identify early epithelial somatic mutations/indels in precancerous breast ducts by comparing genetic DNA sequences from cells obtained from venous blood and ductal lavage | At six months
  Extract high-quality DNA and RNA from human whole blood and ductal lavage (DL) samples. Assess QC and Quantitation of extracted RNA and DNA samples. Assess QC and Quantitation of libraries generated by CGL for Whole Genome DNA-seq and RNA sequencing assays. Sequence prepared libraries using the Illumina Next Generation Sequencing platform.

SECONDARY OUTCOMES:
RNA Sequencing on the Illumina Next Generation Sequencing Platform to identify mRNA hyperplasia or precancerous driver pathways | At six months
  Extract high-quality DNA and RNA from human whole blood and ductal lavage (DL) samples. Assess QC and Quantitation of extracted RNA and DNA samples. Assess QC and Quantitation of libraries generated by CGL for Whole Genome DNA-seq and RNA sequencing assays. Sequence prepared libraries using the Illumina Next Generation Sequencing platform.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Susan Love, MD, Principal Investigator — The Dr. Susan Love Research Foundation
Locations (1):
- Dr. Susan Love Research Foundation, Santa Monica, California, United States

REFERENCES:
- [Background] Mahoney ME, Gordon EJ, Rao JY, Jin Y, Hylton N, Love SM. Intraductal therapy of ductal carcinoma in situ: a presurgery study. Clin Breast Cancer. 2013 Aug;13(4):280-6. doi: 10.1016/j.clbc.2013.02.002. Epub 2013 May 9. PMID 23664819
- [Background] Love SM, Zhang W, Gordon EJ, Rao J, Yang H, Li J, Zhang B, Wang X, Chen G, Zhang B. A feasibility study of the intraductal administration of chemotherapy. Cancer Prev Res (Phila). 2013 Jan;6(1):51-8. doi: 10.1158/1940-6207.CAPR-12-0228. Epub 2012 Nov 20. PMID 23169924
- [Background] Mannello F, Ligi D. Resolving breast cancer heterogeneity by searching reliable protein cancer biomarkers in the breast fluid secretome. BMC Cancer. 2013 Jul 12;13:344. doi: 10.1186/1471-2407-13-344. PMID 23849048
- [Background] Ma CX, Ellis MJ. The Cancer Genome Atlas: clinical applications for breast cancer. Oncology (Williston Park). 2013 Dec;27(12):1263-9, 1274-9. PMID 24624545
- [Background] Kaur H, Mao S, Shah S, Gorski DH, Krawetz SA, Sloane BF, Mattingly RR. Next-generation sequencing: a powerful tool for the discovery of molecular markers in breast ductal carcinoma in situ. Expert Rev Mol Diagn. 2013 Mar;13(2):151-65. doi: 10.1586/erm.13.4. PMID 23477556
- See also: Dr. Susan Love Research Foundation — http://dslrf.org/actwithlove/